CLINICAL TRIAL: NCT06547138
Title: Prospective Descriptive Multicentre Pilot Study On The Effectiveness and Safety Of Optilene® Silver Mesh Elastic In Prevention Of Surgical Site Infection (SSI) And Incisional Hernia (IH)
Brief Title: Pilot Study on the Effectiveness and Safety of OPTILENE® SILVER MESH ELASTIC in Prevention of Surgical Site Infection (SSI) and Incisional Hernia (IH)
Acronym: SSIHLVER
Status: Not yet recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-G-H-2126
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Abdominal Aortic Aneurysm; Morbid Obesity
Keywords: urgent, primary median laparotomy
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Optilene® Silver Mesh Elastic: Prophylactic mesh in high-risk patients
  Interventions: Device: Prophylactic mesh

INTERVENTIONS:
Device: Prophylactic mesh — Prevention of incisional hernia after a prophylactic mesh in high-risk patients

SUMMARY:
The aim of the study is to describe the effectiveness of Optilene® Silver Mesh Elastic on prevention of surgical site infection (SSI) at 6 months follow-up in patients undergoing urgent laparotomy by collecting clinical data on the SSI rates, IH rates and overall clinical performance of Optilene® Silver Mesh Elastic used for the prevention of incisional hernia as prophylactic mesh in patients that require urgent median laparotomy in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Surgical procedure requiring urgent, primary median laparotomy, which are classified as "Class III/Contaminated" or "Class IV/Dirty-Infected" regarding the CDC classification.

These include but are not limited to:

* Vascular surgery
* Colon and rectum
* Hepatobiliary
* Gastrointestinal
* Gynecology
* Urology
* Abdominal Aortic Aneurysm (AAA) repair
* Right hemicolectomy
* Left hemicolectomy
* Sigmoidectomy
* Anterior resection
* Abdominoperineal amputation
* Exploratory laparotomy
* Cholecystectomy
* Cholecystectomy and choledocotomy

  * Written informed consent

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Patients < 18 years old or patients who are still in the growth phase
* Contaminated and infected areas
* Hypersensitivity to silver
* Direct contact with the viscera
* Previous allergic reactions to components of the device
* Patient with previous laparotomy
* Transverse laparotomy
* Patients with previous hernia repair
* Simultaneous participation in another investigational clinical trial (drug or medical studies)
* Patients with active oncologic treatment (chemo and radiotherapy)
* Underlying autoimmune disease
* Recent cardiovascular complication
* Gynecology surgery
* Urology surgery
* Vascular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients according to the professional criteria (such as but not limited to: age, nutrition, body mass index, comorbidities, etc.) who are undergoing prophylactic mesh implantation to avoid surgical site infection after an emergency or urgent intra-abdominal laparotomy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) A2/A3 rate | at 6 months follow-up
  SSIs remain a significant clinical problem as they are associated with substantial mortality and morbidity and impose severe demands on healthcare resources. Centers for Disease Control and Prevention Surgical Site Infection (SSI) Classification System differentiates Superficial SSI (A1), Deep Incisional SSI (A2) and Infection with involvement of organs/body cavities (A3). Only cases of A2 and A3 are considered for the Primary Outcome and are compared to rates from reference literature

SECONDARY OUTCOMES:
Cumulative rate of of postoperative complications during the study period | at discharge (up to 10 days after surgery), 1 month, 6 months, 1 year and 2 year follow-up
  Numbers of all postoperative complications such as mortality, burst abdomen, bowel obstruction, bulging, necrosis, fistula, wound dehiscence, hematoma, seroma, peritonitis are added to the overall complication rate that is observed over the postoperative course
Cumulative Surgical Site Infection (SSI) A2/A3 rate during the study period | at 1 month, 1 year and 2 year follow-up.
  Number of the Surgical Site Infection (SSI) (only A2 and A3) rate at every follow-up
Incisional hernia (IH) rate during the study period | repeatedly at 6 months, 1 year and 2 year follow-up.
  Incisional hernia (IH) is a protrusion of tissue that forms at the site of a healing surgical scar. Incisional hernia refers to abdominal wall hernia at the site of a previous surgical incision.
Length of hospital stay | at discharge (approximately up to 10 days after surgery)
  Number of days the patient has to stay in hospital after the surgery
Development of Pain: Visual Analogue Scale (VAS) | at discharge (approximately up to 10 days after surgery), 1 month, 6 months, 1 year and 2 year follow-up, using the VAS score
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".
Time to return to work | at all postoperative examinations with a single value for each individual patient
  The number of days needed to return to work after the surgery of the individual patient is documented
Handling of the Optilene® Silver Mesh Elastic | intraoperatively
  The handling will be evaluated using a questionnaire (Likert-type scale) with the dimensions Tensile Strength, Absence of memory effect, Elasticity, Stiffness, Surface weight, Thickness, Ease of being fixed with suture, Ease of package extraction as well as an overall opinion in five evaluation levels (excellent=1, very good=2, good=3, satisfied=4, poor=5)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Troyano Escribano, Dr., Principal Investigator — Fundació Hospital de l'Esperit Sant
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Tries i Pujol, Badalona
  - Hospital Municipal Badalona, Badalona
  - Hospital Comarcal Sant Jaume de Calella, Calella
  - Hospital de Mataró, Mataró
  - Hospital Fundació Esperit Sant, Santa Coloma de Gramenet

IPD SHARING:
Plan to Share IPD: No